CLINICAL TRIAL: NCT07301372
Title: A Randomized, Open-label, Blinded Endpoint Evaluation Study of Early Administration of Evolocumab After Thrombolysis in Patients With Atherosclerotic Acute Ischemic Stroke
Brief Title: Evaluation Study of Early Administration of Evolocumab After Thrombolysis in Patients With Atherosclerotic Acute Ischemic Stroke
Acronym: EPOCH-LYSIS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XYFY2025-KL477-02
Record Dates: First submitted 2025-11-27; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Acute Stroke
Keywords: PCSK9 inhibitor; Inflammatory factor; Biomarkers of brain injury; Atorvastatin; Early neurological deterioration
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- evolocumab (Experimental): Within 24 hours after thrombolysis, patients received subcutaneous injections of 420 mg evokine and three vials of evokine, along with standard statin therapy (atorvastatin 20 mg/day).
  Interventions: Drug: Ivolumab 420mg (three vials)
- Standard of care (No Intervention): Following thrombolysis, the patient received standard statin therapy (atorvastatin 20 mg/day).

INTERVENTIONS:
Drug: Ivolumab 420mg (three vials) — Administer 420 mg (three vials) of evolocumab subcutaneously within 24 hours after thrombolysis.
  Arms: evolocumab

SUMMARY:
This study is a Phase IIa clinical trial initiated by the researchers, which is prospective, single-center, randomized, open-label, with blinded endpoint evaluation (PROBE design). Patients were screened through the emergency stroke green channel and included if they had an onset within 9 hours, met the criteria for large artery atherosclerosis (LAA) after multimodal imaging screening, received intravenous thrombolysis, and signed informed consent to participate. The study used block randomization (block size of 4), stratified by baseline National Institutes of Health Stroke Scale (NIHSS) score (5-10 vs >10-20) and onset-to-thrombolysis time (<4.5 hours vs 4.5-9 hours).

Intervention group: received subcutaneous injections of Ilyumumab 420 mg (three syringes) within 24 hours after thrombolysis plus standard drug therapy (including statins). Control group: received conventional statin therapy (atorvastatin 20 mg/day) after thrombolysis. All patients received standardized stroke treatment (initiating antiplatelet therapy 24 hours after thrombolysis) and standardized management of blood pressure and blood glucose.

NIHSS scores were assessed every 12 hours within 72 hours post-thrombolysis, and then daily thereafter, to evaluate the effectiveness of combined therapy in reducing early neurological deterioration (END).

Blinding: The study is open-label. An independent Clinical Endpoint Committee (CEC) was established, and all clinical endpoint events (END assessment, 90-day mRS scores) were evaluated in a blinded manner by experts who were completely unaware of group assignments.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-85 years. No gender or sex restrictions, and no gender ratio restrictions.

2. Clinically diagnosed with acute ischemic stroke, with the time from symptom onset to intravenous thrombolysis <9 hours.

1. Within 4.5 hours of symptom onset: This time window is based on the ECASS III criteria (Class IA recommendation) and is currently the standard indication for intravenous thrombolysis in acute ischemic stroke worldwide.
2. 4.5-9 hours: Referring to the EXTEND study criteria, meeting the following multimodal imaging mismatch ratio: ischemic penumbra volume/ischemic core volume >1.2, with an absolute mismatch volume >10 mL and an ischemic core volume <70 mL.

3. The stroke meets the TOAST classification for large artery atherosclerosis (LAA), which includes intracranial arteriosclerosis (ICAS) and extracranial arteriosclerosis (ECAS), and meets one of the following three criteria: large artery stenosis ≥50%, infarct lesion >1.5cm + ipsilateral plaque (no stenosis requirement), or intracranial artery stenosis ≥30% with plaque ulceration.

4. The patient or their legal representative has signed an informed consent form.

Exclusion Criteria:

1. CT scan showing signs of intracranial hemorrhage, symptomatic intracranial hemorrhage, or subarachnoid hemorrhage, even if the CT scan results are normal.

2. Patients who must or wish to continue using restrictive medications or any medications that may interfere with the safe conduct of the trial.

3. Acute bleeding tendency, including but not limited to:

1. A known family history of bleeding disorders and a history of a serious bleeding disorder currently present or within the past 6 months.
2. Receiving heparin treatment within the past 48 hours, with an activated partial thromboplastin time (aPTT) exceeding the upper limit of the normal range for laboratory testing.
3. Currently taking an oral vitamin K anticoagulant (e.g., warfarin) with a prolonged prothrombin time (INR > 1.7 or PT > 15 seconds); or currently taking a novel oral anticoagulant (e.g., dabigatran etexilate, rivaroxaban, or apixaban) with an activated partial thromboplastin time (aPTT) and/or prothrombin time (PT) exceeding the upper limit of the local laboratory reference range.
4. Platelet count below 100,000/mm³ at screening.
5. History of central nervous system injury (e.g., tumor, aneurysm, intracranial or spinal surgery).
6. Experiencing traumatic external cardiac compression, obstetric delivery, or non-compressive vascular puncture (e.g., subclavian or jugular vein puncture) within the past 10 days.
7. Known history of suspected intracranial hemorrhage or suspected aneurysm/subarachnoid hemorrhage.
8. Tumors with increased bleeding risk.
9. History of ulcerative gastrointestinal disease, esophageal varices, aneurysm, or arteriovenous malformation within the past 3 months.
10. Associated with bleeding risk. 4. Any known disease significantly associated with this condition.

4. Previous mRS score ≥2, with comorbid dementia or other neurodegenerative diseases.

5. Clinically confirmed non-atherosclerotic intracranial arterial stenosis, such as aortic dissection, vasculitis, moyamoya disease, embolism, immune system disorders, etc.

6. Other comorbid medical histories that may affect endpoint event determination and follow-up, such as history of traumatic brain injury, multiple sclerosis, encephalitis, tumors, poisoning, syphilis, and severe heart, lung, liver, kidney, or endocrine diseases.

7. Pregnant women.

8. Currently participating in other experimental device or drug studies, or having completed other experimental device or drug studies, or having received other experimental treatments for less than 30 days.

9. Having used PCSK9 inhibitors within 4 weeks prior to enrollment.

10. Hypersensitivity to statins or PCSK9 inhibitors.

11. Patients with severe hepatic or renal impairment (eGFR <30 ml/min/1.73 m²).

12. Refusal to sign informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Early deterioration of neurological function (END) | within 1-7 days after thrombolysis.
  Defined as an increase of ≥2 points in NIHSS score or death within 1-7 days after thrombolysis. NIHSS scores should be assessed daily.The NIHSS (National Institutes of Health Stroke Scale) has a total score of 0 to 42. The higher the total score, the more severe the neurological deficit caused by stroke.

SECONDARY OUTCOMES:
Therapeutic efficacy | Within 90 days after thrombolysis
  90-day functional prognosis (mRS 0-2 score rate and ordered shift analysis).The Modified Rankin Scale (MRS) is a core tool for assessing the degree of neurological function recovery in patients with stroke or other neurological disorders. The score ranges from 0 to 6, with higher scores indicating a more severe degree of disability.
Mechanism exploration | from baseline to 36 hours and 72 hours after thrombolysis.
  Dynamic changes in serum PCSK9 levels from baseline to 36 hours and 72 hours after thrombolysis,and the correlation between these changes and the end of the treatment period.
Mechanism Exploration | from baseline to 36 hours and 72 hours after thrombolysis
  Dynamic changes in serum hsCRP levels from baseline to 36 hours and 72 hours after thrombolysis,and the correlation between these changes and the end of the treatment period.
Mechanism Exploration | from baseline to 36 hours and 72 hours after thrombolysis
  Dynamic changes in serum IL-6 levels from baseline to 36 hours and 72 hours after thrombolysis,and the correlation between these changes and the end of the treatment period.
Mechanism Exploration | from baseline to 36 hours and 72 hours after thrombolysis
  Dynamic changes in serum NSE and S100β levels from baseline to 36 hours and 72 hours after thrombolysis, and the correlation between these changes and the end of the treatment period.
Preset subgroup analysis | within 1-7 days after thrombolysis
  The impact of onset to thrombolysis time (<4.5h vs 4.5-9h) on the primary efficacy endpoint.The efficacy therapeutic endpoint was early deterioration of neurological function (END).Defined as an increase of ≥2 points in NIHSS score or death within 1-7 days after thrombolysis. NIHSS scores should be assessed daily.The NIHSS (National Institutes of Health Stroke Scale) has a total score of 0 to 42. The higher the total score, the more severe the neurological deficit caused by stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Ren Guo Chen, Study Director — the Ethics Committee of the Affiliated Hospital of Xuzhou Medical University
Locations (1):
- Department of Neurology, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Participants do not consent to the data sharing about themselves. IPD involves privacy and ethical issues.